CLINICAL TRIAL: NCT00743431
Title: Caelyx in Ovarian Cancer: Prevention and Treatment of Infusion Reactions and Palmar-plantar Erythrodysesthesia (PPE).
Brief Title: Caelyx in Ovarian Cancer: Prevention and Treatment of Infusion Reactions and Palmar-plantar Erythrodysesthesia (Study P04085)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04085
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women with advanced ovarian cancer
  Interventions: Drug: Caelyx (Pegylated Lyposomal Doxorubicin)

INTERVENTIONS:
Drug: Caelyx (Pegylated Lyposomal Doxorubicin) — Pegylated Lyposomal Doxorubicin, 50 mg/m2 every 4 weeks for 6 cycles.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Caelyx in women with advanced ovarian cancer, focusing on infusion reactions and palmar-plantar erythrodysesthesia.

DETAILED DESCRIPTION:
This observational program is aimed at gaining tolerability and safety data with the routine use of Caelyx in its labelled indication in ovarian cancer, focusing on infusion reaction and PPE.

Data will be raised about the premedication routinely used for the prevention of side effects caused by Caelyx. Premedications for infusion reactions include corticosteroids, serotonin 3 (5HT3) antagonists, histamine 1 (H1) blockers, and histamine 2 (H2) blockers. Premedications for PPE include oral dexamethasone and vitamin B6.

The management of infusion reactions and PPE will be recorded. A detailed record of the medical history may reveal patient groups at a higher risk of experiencing these side effects.

ELIGIBILITY:
Inclusion Criteria:

* Women with advanced ovarian cancer with:

  * previous platin/taxane therapy and documented measureable and/or evaluable advanced or metastatic cancer by radiological imaging or increase of serum cancer antigen 125 (CA 125) according to Rustin et al.

Exclusion Criteria:

* Patients that are not treated according to the Austrian Summary of Product Characteristics (SPC)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with advanced ovarian cancer with:
  previous platin/taxane therapy and
  documented measurable and/or evaluable advanced or metastatic cancer by radiological imaging or increase of serum cancer antigen 125 (CA 125) according to Rustin et al.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Result] Steppan I, Reimer D, Sevelda U, Ulmer H, Marth C, Zeimet AG. Treatment of recurrent platinum-resistant ovarian cancer with pegylated liposomal doxorubicin--an evaluation of the therapeutic index with special emphasis on cardiac toxicity. Chemotherapy. 2009;55(6):391-8. doi: 10.1159/000262452. Epub 2009 Nov 30. PMID 19955744

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated Lyposomal Doxorubicin: 50 mg/m2 every 4 weeks for 6 cycles
Period: Overall Study
Arm/Group | Pegylated Lyposomal Doxorubicin
Started | 224
Completed | 98
Not Completed | 126
Not completed — Toxicity | 6
Not completed — Tumor progression | 56
Not completed — Withdrawal by Subject | 13
Not completed — Death | 9
Not completed — Reason for discontinuation not specified | 29
Not completed — No documentation available | 13

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated Lyposomal Doxorubicin
Number analyzed (Participants) | 224
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age was calculated for the Intent-to-Treat (ITT) population of 214.
  years | 62.4 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 0
Region of Enrollment [Number; unit: participants]
  Austria | 224

OUTCOME MEASURES:

1. Primary Outcome: Occurrences of Infusion Reactions and Palmar-Plantar Erythrodysesthesia (PPE)
Description: Definitions in assessment of adverse event severity:
  Mild: awareness of sign, symptom, or event, but easily
  tolerated.
  Moderate: discomfort enough to cause interference with usual
  activity and may warrant intervention.
  Severe: incapacitating with inability to do usual activities or
  significantly affects clinical status, and warrants
  intervention.
Time Frame: The observational program was conducted over a period of 2 years
Population: Intent-to-treat (ITT) (N=214). This is also the Safety population.
Measure: Number; unit: Events
Arm/Group | Pegylated Lyposomal Doxorubicin
Number analyzed (Participants) | 214
Events
  Mild infusion reaction | 2
  Moderate infusion reaction | 5
  Severe infusion reaction | 2
  infusion reaction - severity not specified | 1
  Mild PPE | 37
  Moderate PPE | 23
  Severe PPE | 5

ADVERSE EVENTS:
Description: Population of 214 was the Safety population as well as the Intent-to-Treat (ITT) population.
Arm/Group | Pegylated Lyposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 14/214
Other Adverse Events (participants affected / at risk) | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Lyposomal Doxorubicin (N=214)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
General physical health deterioraton (General disorders) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No